CLINICAL TRIAL: NCT04550494
Title: A Pharmacodynamics-Driven Trial of Talazoparib, an Oral PARP Inhibitor, in Patients With Advanced Solid Tumors and Aberrations in Genes Involved in DNA Damage Response
Brief Title: Measuring the Effects of Talazoparib in Patients With Advanced Cancer and DNA Repair Variations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-06906; NCI-2020-06906 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 000264; 000246; 10371 (Other: National Cancer Institute LAO); 10371 (Other: CTEP); NCT04692662 (obsolete NCT alias)
Record Dates: First submitted 2020-09-15; First posted 2020-09-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Castration-Resistant Prostate Carcinoma; Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage IV Gastric Cancer AJCC v8; HER2-Positive Breast Carcinoma; Locally Advanced Breast Carcinoma; Locally Advanced Gastric Carcinoma; Locally Advanced Malignant Solid Neoplasm; Locally Advanced Ovarian Carcinoma; Locally Advanced Pancreatic Carcinoma; Locally Advanced Prostate Carcinoma; Metastatic Breast Carcinoma; Metastatic Gastric Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Ovarian Carcinoma; Metastatic Pancreatic Carcinoma; Metastatic Prostate Carcinoma; Platinum-Sensitive Ovarian Carcinoma; Recurrent Breast Carcinoma; Recurrent Gastric Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Pancreatic Carcinoma; Recurrent Prostate Carcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Neoplasm Metastasis; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (talazoparib) (Experimental): Patients receive talazoparib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo biopsy and blood sample collection as well as CT scan or MRI throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Talazoparib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Talazoparib — Given PO
  Other Names: BMN 673; BMN-673; BMN673

SUMMARY:
This phase II trial studies if talazoparib works in patients with cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) and has mutation(s) in deoxyribonucleic acid (DNA) damage response genes who have or have not already been treated with another PARP inhibitor. Talazoparib is an inhibitor of PARP, a protein that helps repair damaged DNA. Blocking PARP may help keep cancer cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. All patients who take part on this study must have a gene aberration that changes how their tumors are able to repair DNA. This trial may help scientists learn whether some patients might benefit from taking different PARP inhibitors "one after the other" and learn how talazoparib works in treating patients with advanced cancer who have aberration in DNA repair genes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the pharmacodynamic (PD) effect of talazoparib in tumor biopsies for patients with aberrations in deoxyribonucleic acid (DNA) damage response genes who have or have not received prior PARP inhibitor treatment (separately).

SECONDARY OBJECTIVE:

I. Determine the response rate (complete response [CR] + partial response [PR]) of treatment with talazoparib in patients with aberrations in DNA damage response genes.

EXPLORATORY OBJECTIVE:

I. Investigate tumor genomic alterations potentially associated with sensitivity or acquired resistance to talazoparib.

OUTLINE:

Patients receive talazoparib orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo biopsy and blood sample collection, as well as computed tomography (CT) scan or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with solid tumors and documented germline or somatic aberrations in genes involved in DNA damage response (DDR) and whose disease has progressed following at least one standard therapy or who have no acceptable standard treatment options. Molecular testing performed at an National Cancer Institute-Molecular Analysis for Therapy Choice (NCI-MATCH) (NCT02465060) study-designated Clinical Laboratory Improvement Act (CLIA) laboratory or at Myriad Genetics, GeneDx, Invitae, or the Frederick National Laboratory for Cancer Research (FNLCR) Molecular Characterization Laboratory (MoCha) will be acceptable for determination of eligibility
* Patients with the following germline or somatic genetic aberrations will be eligible based on compelling preclinical and/or clinical data suggesting that these deleterious mutations confer sensitivity to PARP inhibitors; no more than 6 patients (across both cohorts) with an eligibility mutation in any one gene will be enrolled

  * Deleterious BRCA1 or BRCA2 mutations
  * Loss of function mutations (including novel loss of function frameshift or nonsense mutations) in the following Fanconi anemia genes: FANCA, FANCB, FANCC, FANCD2, FANCE, FANCF, FANCG, FANCI, FANCJ, FANCL, FANCM, FANCN
  * A known functional mutation (including novel loss of function frameshift or nonsense mutations) in any of the following DDR genes: ARID1A, ATM, ATR, BACH1 (BRIP1), BAP1, BARD1, CDK12, CHK1, CHK2, IDH1, IDH2, MRE11A, NBN, PALB2, RAD50, RAD51, RAD51B, RAD51C, RAD51D, RAD54L
* Age >= 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 10 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (=< 3 x upper limit of normal in the presence of documented Gilbert's syndrome or liver metastases at baseline)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x institutional upper limit of normal
* Creatinine =< 1.5 x institutional upper limit of normal OR Creatinine clearance (CrCl) >= 60 mL/min/1.73m^2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73m^2
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with CT scan, MRI, or calipers by clinical exam
* Patients must have a tumor site amenable to biopsy. If avoidable, the lesion for biopsy should not be selected as a target lesion for RECIST measurements
* The effects of talazoparib on the developing human fetus are unknown. For this reason and because PARP inhibitors are known to be teratogenic, women of child-bearing potential must agree to use a highly effective method of contraception for the duration of study participation and for at least 7 months after completing study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Male patients with female partners of reproductive potential and pregnant partners who are treated or enrolled on this protocol must also agree to use adequate contraception for the duration of study participation and for at least 4 months after completion of talazoparib administration
* Patients must be able to swallow whole tablets or capsules. Nasogastric or gastric-tube (G-tube) administration is not allowed. Any gastrointestinal disease which would impair ability to swallow, retain, or absorb drug is not allowed
* Ability to understand and the willingness to sign a written informed consent document
* Patients must have recurrent, locally advanced or metastatic disease
* Patients must have progressed on or after at least one line of standard-of-care (SOC) intervention, except for those patients without SOC or for whom talazoparib is SOC
* PATIENTS WITH OVARIAN CANCER:
* All patients with ovarian cancer should have one prior platinum-based therapy
* Patients with ovarian cancer with platinum-sensitive disease are eligible. Patients with platinum-refractory disease are not eligible
* Patients with gBRCAm ovarian cancer must also have progressed on a PARP inhibitor. The time and treatment between the prior PARP inhibitor and protocol initiation must be documented
* PATIENTS WITH PANCREATIC CANCER:
* All patients with pancreatic cancer should have received prior platinum-containing therapy in the metastatic setting
* PATIENTS WITH BREAST CANCER:
* Patients with HER2+ breast cancer should have had 2 prior systemic lines of therapy in the metastatic setting, including anti-HER2 therapy
* Patients with breast cancer who are eligible for a PARP inhibitor by Food and Drug Association (FDA) approvals must have had prior PARP inhibitor as per FDA indication. The time and treatment between the prior PARP inhibitor and protocol initiation must be documented
* PATIENTS WITH GASTRIC CANCER:
* Patients with HER2+ gastric cancer should have had received anti-HER2 therapy in the metastatic setting
* PATIENTS WITH PROSTATE CANCER:
* Patients with prostate cancer who are eligible for a PARP inhibitor by FDA approvals must have had prior PARP inhibitor for eligibility. The time and treatment between the prior PARP inhibitor and protocol initiation must be documented
* All patients with prostate cancer can continue to receive treatment with gonadotropin-releasing hormone (GnRH) agonists while on study, as long as there is evidence of disease progression on prior therapy
* Patients with castration resistant prostate cancer must have castrate levels of testosterone (< 50 ng/dL [1.74 nmol/L])
* Patients with metastatic hormone receptor (HR) prostate cancer and mutations in either BRCA1, BRCA2, or ATM should continue to receive anti-androgen receptor (anti-AR) therapy

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks or 5 half-lives, whichever is shorter (6 weeks for nitrosoureas or mitomycin C). Patients must be >= 2 weeks since any prior administration of a study drug in a phase 0 or equivalent study and be >= 1 week from palliative radiation therapy. Patients must have recovered to eligibility levels from prior toxicity or adverse events
* Patients who have had prior treatment with talazoparib are ineligible
* Patients who have had prior monoclonal antibody therapy must have completed that therapy >= 6 weeks (or 3 half-lives of the antibody, whichever is shorter) prior to enrollment on protocol (minimum of 1 week between prior therapy and study enrollment) except for monoclonal antibody therapies that have been proven to be safe when combined with PARP inhibitor (PARPi) treatment (such as anti-PD-1/PD-L1 and anti-HER2), which must be completed >= 4 weeks prior to enrollment
* Patients who are receiving any other investigational agents
* Patients with active brain metastases or carcinomatous meningitis are excluded from this clinical trial. Patients with treated brain metastases, whose brain metastatic disease has remained stable for >= 1 month without requiring steroid and anti-seizure medication are eligible to participate
* Eligibility of subjects receiving any medications or substances with the potential to affect the activity or pharmacokinetics of talazoparib will be determined following review by the principal investigator
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because the effects of the study drugs on the developing fetus are unknown
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Patients who require use of coumarin-derivative anticoagulants such as warfarin are excluded. Low-dose warfarin (=< 1 mg/day) is permitted
* Women who are currently lactating
* History of prior malignancies within the past 3 years other than non-melanomatous skin cancers that have been controlled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent of patients who demonstrate simultaneous Rad51 activation | At cycle 2 day 1
  Will be measured as the percent of patients who demonstrate simultaneous Rad51 activation, defined to be at least 5% cells with at least 5 Rad51 foci, and lack of gamma-H2AX activation, defined to be less than 4% nuclear area positive (NAP), at the cycle 2 day 1 biopsy.

SECONDARY OUTCOMES:
Overall response rate | Up to 30 days after last dose
  Will estimate the overall response rate (complete response + partial response) among eligible patients who have received at least one dose of talazoparib. A 95% confidence interval for this response rate will also be computed. For this analysis, response classifications will follow Response Evaluation Criteria in Solid Tumors version 1.1 guidelines.

OTHER OUTCOMES:
Tumor genomic alterations potentially associated with sensitivity or acquired resistance to talazoparib | Up to 30 days after last dose
  Exploratory evaluations will be performed, with results reported with appropriate caveats about the exploratory nature of the analysis, and without formal adjustment for multiple comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: A P Chen, Principal Investigator — National Cancer Institute LAO
Locations (4):
- United States (4):
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm